CLINICAL TRIAL: NCT04745715
Title: Genomic Analysis in Surgically Treated NSCLC Brain Metastasis Based on Neurosurgical Perspectives
Brief Title: Genomic Study in Non-small Cell Lung Cancer Brain Metastasis
Status: Completed | Type: Observational
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: A-ER-109-437
Record Dates: First submitted 2021-02-03; First posted 2021-02-09 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2020-12

CONDITIONS: NSCLC Stage IV; Brain Metastases
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Brain Neoplasms | interventions — Craniotomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: craniectomy — craniectomy outcomes and survival

SUMMARY:
The investigators collected the data from the investigators' center between January 2011 and October 2020. The study included all non-small cell lung cancer patients with surgically excised brain metastasis. The investigators analysis the correlation of gene mutation and the disease course.

DETAILED DESCRIPTION:
The investigators collected the data from from the investigators' center between January 2011 and October 2020. The study included all non-small cell lung cancer patients with surgically excised brain metastasis. The investigators analysis the correlation of gene mutation and the disease course. The investigators use Kaplan-Meier regression to analyze the overall survival, and the difference between the groups was calculated using log rank test. Cox proportional hazards method was used to create the regression model and estimate the hazard ratios.

ELIGIBILITY:
Inclusion Criteria:

- patients diagnosed with non-small cell lung cancer who underwent craniectomy and subsequent whole brain radiotherapy and associated chemo or target therapy

Exclusion Criteria:

* patient who did not receive postoperative adjuvant therapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with non-small cell lung cancer underwent craniectomy, who completed postoperative whole brain radiotherapy and associated chemo or target therapy
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
postoperative survival | From date of craniectomy until the date of patient deceased or date of last followed medical record, with median follow up around to 20 months

CONTACTS AND LOCATIONS:
Locations (1):
- National Cheng Kung University hospital, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No